CLINICAL TRIAL: NCT01952145
Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide Versus Insulin Glargine in Subjects With Type 2 Diabetes Mellitus (DUAL™ V - Basal Insulin Switch)
Brief Title: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide Versus Insulin Glargine in Subjects With Type 2 Diabetes Mellitus
Acronym: DUAL™ V
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-3952; 2012-004413-14 (EudraCT Number); U1111-1135-1003 (Other: WHO)
Record Dates: First submitted 2013-09-24; First posted 2013-09-27 (Estimated); Results first posted 2017-01-20 (Estimated); Last update posted 2019-01-03 (Actual); Status verified 2018-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin degludec/liraglutide OD plus metformin (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Insulin glargine OD plus metformin (Active Comparator)
  Interventions: Drug: insulin glargine

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Insulin degludec/liraglutide is injected subcutaneously s.c. (under the skin) once daily (OD). Dose individually adjusted. Subjects should continue their pre-trial treatment with metformin.
  Arms: Insulin degludec/liraglutide OD plus metformin
Drug: insulin glargine — Insulin glargine is injected subcutaneously s.c. (under the skin) once daily (OD). Dose individually adjusted. Subjects should continue their pre-trial treatment with metformin.
  Arms: Insulin glargine OD plus metformin

SUMMARY:
This trial is conducted globally. The aim of the trial is to compare the efficacy and safety of insulin degludec/liraglutide versus insulin glargine in subjects with type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: - Type 2 diabetes mellitus - HbA1c 7.0-10.0% [53-86 mmol/mol] (both inclusive) by central laboratory analysis - Current treatment with insulin glargine for at least 90 days prior to screening - Stable daily dose of insulin glargine between 20 units and 50 units (both inclusive) for at least 56 days prior to screening. Total daily dose should be within the range of 20-50 units, both inclusive, on the day of screening, but individual fluctuations of plus/minus 10 procent within the 56 days prior to screening are acceptable - Stable daily dose of metformin (above or equal to 1500 mg or max tolerated dose) for at least 90 days prior to screening - Body mass index (BMI) below or equal to 40 kg/m^2 Exclusion Criteria: - Any use of oral antidiabetic agents (OADs) (except for metformin) within 90 days prior to Visit 1 (screening) - Current use of any drug (except metformin and insulin glargine) or anticipated change inconcomitant medication, which in the investigator's opinion could interfere with the glucose metabolism (e.g. systemic corticosteroids) - Previous and/or current treatment with any insulin regimen other than basal insulin, e.g. prandial or pre-mixed insulin (short term treatment due to intercurrent illness includinggestational diabetes is allowed at the discretion of the investigator) - Previous and/or current treatment with glucagon-like peptide-1 (GLP-1) receptor agonists (e.g. exenatide, liraglutide) - Impaired liver function, defined as ALAT (alanine aminotransferase) above or equal to 2.5 times upper normal range (UNR) - Impaired renal function defined as serum-creatinine above or equal to 133 micromol/L (above or equal to 1.5 mg/dL) for males and above or equal to 125 micromol/L (1.4 mg/dL) for females, or as allowed according to local contraindications for metformin - Screening calcitonin above or equal to 50 ng/L - Personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN2) - History of chronic pancreatitis or idiopathic acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2014-11-04 (Actual); Study Completion 2014-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (80):
- United States (29):
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Los Alamitos, California
  - Novo Nordisk Investigational Site, Palm Springs, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, Evansville, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Louisville, Kentucky
  - Novo Nordisk Investigational Site, Slidell, Louisiana
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Wilmington, North Carolina
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Altoona, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Collierville, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, West Jordan, Utah
  - Novo Nordisk Investigational Site, Renton, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
- Argentina (5):
  - Novo Nordisk Investigational Site, Buenos Aires
  - Novo Nordisk Investigational Site, Capital Federal
  - Novo Nordisk Investigational Site, Corrientes
  - Novo Nordisk Investigational Site, Salta
  - Novo Nordisk Investigational Site, Zárate
- Australia (6):
  - Novo Nordisk Investigational Site, Blacktown, New South Wales
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, Herston, Queensland
  - Novo Nordisk Investigational Site, Ipswich, Queensland
  - Novo Nordisk Investigational Site, Robina, Queensland
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
- Greece (4):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Thessaloniki
- Hungary (5):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Győr
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Miskolc
- Mexico (5):
  - Novo Nordisk Investigational Site, Pachuca, Hidalgo
  - Novo Nordisk Investigational Site, Cuernavaca, Morelos
  - Novo Nordisk Investigational Site, Mexico City, México, D.F.
  - Novo Nordisk Investigational Site, Durango
  - Novo Nordisk Investigational Site, Monterrey
- Russia (8):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Kirov
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Volgograd
  - Novo Nordisk Investigational Site, Vsevolozhsk
- Slovakia (10):
  - Novo Nordisk Investigational Site, Bardejov
  - Novo Nordisk Investigational Site, Dolný Kubín
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Levice
  - Novo Nordisk Investigational Site, Ľubochňa
  - Novo Nordisk Investigational Site, Poprad
  - Novo Nordisk Investigational Site, Považská Bystrica
  - Novo Nordisk Investigational Site, Prievidza
  - Novo Nordisk Investigational Site, Trnava
  - Novo Nordisk Investigational Site, Veľký Meder
- South Africa (3):
  - Novo Nordisk Investigational Site, Midrand, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Alberton
- Spain (5):
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Palma de Mallorca
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia

REFERENCES:
- [Result] Lingvay I, Perez Manghi F, Garcia-Hernandez P, Norwood P, Lehmann L, Tarp-Johansen MJ, Buse JB; DUAL V Investigators. Effect of Insulin Glargine Up-titration vs Insulin Degludec/Liraglutide on Glycated Hemoglobin Levels in Patients With Uncontrolled Type 2 Diabetes: The DUAL V Randomized Clinical Trial. JAMA. 2016 Mar 1;315(9):898-907. doi: 10.1001/jama.2016.1252. PMID 26934259
- [Result] Hunt B, Mocarski M, Valentine WJ, Langer J. Evaluation of the long-term cost-effectiveness of IDegLira versus liraglutide added to basal insulin for patients with type 2 diabetes failing to achieve glycemic control on basal insulin in the USA. J Med Econ. 2017 Jul;20(7):663-670. doi: 10.1080/13696998.2017.1301943. Epub 2017 Mar 15. PMID 28294641
- [Result] Hunt B, Mocarski M, Valentine WJ, Langer J. Evaluation of the Short-Term Cost-Effectiveness of IDegLira Versus Continued Up-Titration of Insulin Glargine U100 in Patients with Type 2 Diabetes in the USA. Adv Ther. 2017 Apr;34(4):954-965. doi: 10.1007/s12325-017-0502-2. Epub 2017 Mar 9. PMID 28281218
- [Result] Norwood P, Chen R, Jaeckel E, Lingvay I, Jarlov H, Lehmann L, Heller S. Rates of hypoglycaemia are lower in patients treated with insulin degludec/liraglutide (IDegLira) than with IDeg or insulin glargine, regardless of the hypoglycaemia definition used. Diabetes Obes Metab. 2017 Nov;19(11):1562-1569. doi: 10.1111/dom.12972. Epub 2017 Jul 10. PMID 28417535
- [Result] Lingvay I, Harris S, Jaeckel E, Chandarana K, Ranthe MF, Jodar E. Insulin degludec/liraglutide (IDegLira) was effective across a range of dysglycaemia and body mass index categories in the DUAL V randomized trial. Diabetes Obes Metab. 2018 Jan;20(1):200-205. doi: 10.1111/dom.13043. Epub 2017 Jul 31. PMID 28643425
- [Result] Psota M, Psenkova MB, Racekova N, Ramirez de Arellano A, Vandebrouck T, Hunt B. Cost-effectiveness analysis of IDegLira versus basal-bolus insulin for patients with type 2 diabetes in the Slovak health system. Clinicoecon Outcomes Res. 2017 Dec 12;9:749-762. doi: 10.2147/CEOR.S143127. eCollection 2017. PMID 29276398
- [Result] Lingvay I, Handelsman Y, Linjawi S, Vilsboll T, Halladin N, Ranc K, Liebl A. EFFICACY AND SAFETY OF IDEGLIRA IN OLDER PATIENTS WITH TYPE 2 DIABETES. Endocr Pract. 2019 Feb;25(2):144-155. doi: 10.4158/EP-2018-0284. Epub 2018 Nov 1. PMID 30383495
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- [Derived] Philis-Tsimikas A, Aroda VR, De Block C, Billings LK, Liebl A, Sivarathinasami R, D'Cruz JM, Lingvay I. Higher Derived Time in Range With IDegLira Versus Insulin Glargine U100 in People With Type 2 Diabetes. J Diabetes Sci Technol. 2024 May;18(3):653-659. doi: 10.1177/19322968221149041. Epub 2023 Jan 29. PMID 36710452
- [Derived] Meneghini L, Doshi A, Gouet D, Vilsboll T, Begtrup K, Orsy P, Ranthe MF, Lingvay I. Insulin degludec/liraglutide (IDegLira) maintains glycaemic control and improves clinical outcomes, regardless of pre-trial insulin dose, in people with type 2 diabetes that is uncontrolled on basal insulin. Diabet Med. 2020 Feb;37(2):267-276. doi: 10.1111/dme.14178. Epub 2019 Nov 28. PMID 31705547
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 75 sites in 10 countries as follows: Argentina: 5 sites; Australia: 4 sites; Greece: 6 sites, Hungary: 4 sites; Mexico: 5 sites, Russian Federation: 11 sites; Slovakia: 11 sites, South Africa: 4 sites; Spain: 6 sites, United States: 19 sites.
Pre-assignment Details: Subjects who were recruited had T2DM and were required to have been on treatment with stable daily dose of insulin glargine between 20 units and 50 units (both inclusive) for at least 56 days prior to screening in combination with a stable daily dose of metformin (≥1500 mg or max tolerated dose) for at least 90 days prior to screening.
Groups:
- Insulin Degludec/Liraglutide (IDegLira): Eligible subjects received IDegLira once daily (OD) subcutaneously for a duration of 26 weeks. The starting dose of IDegLira was 16 dose steps (16 units IDeg/0.6 mg liraglutide) and was titrated according to a predefined titration algorithm with a maximum dose of 50 dose steps (50 units IDeg/1.8 mg liraglutide). Adjustment of the dose was performed twice weekly based on the mean of 3 preceding daily fasting SMPG values on 3 consecutive days. Adjustments were made in increments or decrements of 2 dose steps, aiming at a fasting glycaemic target of 4.0-5.0 mmol/L (71-90 mg/dL). That is, the adjustments were +2 or -2 if the mean of 3 pre-breakfast SMPG values were >5.0 mmol/L (or >90 mg/dL) and <4.0 mmol/L (or <71 mg/dL) respectively. No adjustment was done when the mean of 3 pre-breakfast SMPG values were 4.0 - 5.0 mmol/L (or 71-90 mg/dL). The subjects continued with pre-trial doses of metformin, unless there was a safety concern.
- Insulin Glargine (IGlar): Eligible subjects received IGlar OD subcutaneously for a duration of 26 weeks. The treatment started with dose equal to the pre-trial daily dose (dose-to-dose switch), after which the dose was titrated according to the specified titration algorithm aiming at a fasting glycaemic target of 4.0-5.0 mmol/L (71-90 mg/dL). No predefined maximum dose was specified for IGlar. The subjects continued with pre-trial doses of metformin, unless there was a safety concern.
Period: Overall Study
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar)
Started | 278 | 279
Completed | 250 | 265
Not Completed | 28 | 14
Not completed — Protocol Violation | 2 | 1
Not completed — Death | 0 | 1
Not completed — Adverse Event | 9 | 0
Not completed — Withdrawal Criteria | 16 | 11
Not completed — Unclassified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was used for baseline measurements. FAS included all randomised subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar) | Total
Number analyzed (Participants) | 278 | 279 | 557
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.4 (9.8) | 59.1 (9.3) | 58.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 135 | 142 | 277
  Male | 143 | 137 | 280
Glycated hemoglobin (HbA1c) [Mean (Standard Deviation); unit: Percentage (%)] | 8.4 (0.9) | 8.2 (0.9) | 8.3 (0.9)
Body weight [Mean (Standard Deviation); unit: Kg] | 88.3 (17.5) | 87.3 (15.8) | 87.8 (16.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Haemoglobin)
Description: Change from baseline in HbA1c after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: FAS was used for analysis of this endpoint. And FAS included all randomised subjects. Missing values (including intermittent missing values) were imputed using the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 278 | 279
Percentage (%) | -1.81 (1.08) | -1.13 (0.98)
Statistical Analysis 1: Comparison: Insulin Degludec/Liraglutide (IDegLira) vs Insulin Glargine (IGlar); This primary endpoint was analysed on the FAS using an ANCOVA model with treatment and region as fixed effects and baseline HbA1c value as covariate; Test type: Non-Inferiority or Equivalence — Non-inferiority of IDegLira versus IGlar was considered as confirmed, if the 95% confidence interval (CI) for the mean treatment difference was entirely below 0.30%; p < 0.001, ANCOVA; Treatment contrast = -0.59, 95% CI 2-sided [-0.74 to -0.45]

2. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight after 26 weeks of treatment
Time Frame: Week 0, week 26
Population: FAS which included all randomised subjects was used for analysis of this endpoint. Missing values (including intermittent missing values) were imputed using LOCF method.
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 278 | 279
Kg | -1.4 (3.5) | 1.8 (3.6)

3. Secondary Outcome: Number of Treatment Emergent Confirmed Hypoglycaemic Episodes
Description: Confirmed hypoglycaemic episodes were defined as either: Severe (i.e., an episode requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions) or an episode biochemically confirmed by a plasma glucose value of <3.1 mmol/L (56 mg/dL), with or without symptoms consistent with hypoglycaemia.
Time Frame: During 26 weeks of treatment
Population: The safety analysis set was used for analysis of this endpoint and this set included all subjects receiving at least one dose of trial product. Subjects contributed to the evaluation "as treated". Confirmed hypoglycaemic episodes were reported by 79 subjects in IdegLira arm and by 137 subjects in IGlar arm.
Measure: Number; unit: Number of episodes
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar)
Number analyzed (Participants) | 278 | 279
Number of episodes | 289 | 683

ADVERSE EVENTS:
Time Frame: Week 0 to week 27 (26-week treatment period and a follow-up visit 1 week after end of treatment)
Description: All AEs described below are treatment-emergent. A treatment-emergent AE (TEAE) was defined as an event that had onset date on or after the first day of exposure to randomised treatment and no later than 7 days after the last day of randomised treatment. Analysis population: safety analysis set.
Arm/Group | Insulin Degludec/Liraglutide (IDegLira) | Insulin Glargine (IGlar)
Serious Adverse Events (participants affected / at risk) | 5/278 | 9/279
Other Adverse Events (participants affected / at risk) | 52/278 | 22/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (IDegLira) (N=278) | Insulin Glargine (IGlar) (N=279)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Auricular perichondritis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Degludec/Liraglutide (IDegLira) (N=278) | Insulin Glargine (IGlar) (N=279)
Diarrhoea (Gastrointestinal disorders) | 20 (23) | 7 (10)
Headache (Nervous system disorders) | 11 (12) | 14 (28)
Nausea (Gastrointestinal disorders) | 26 (34) | 3 (3)
Vomiting (Gastrointestinal disorders) | 14 (22) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.